CLINICAL TRIAL: NCT03303807
Title: Study of Carbon Dioxide Removal to Alleviate Right Ventricule Dysfunction During Acute Respiratory Distress Syndrome
Brief Title: Correction by ECCO2-R of Hypercapnia in Patients With DVP in Moderate to Severe ARDS Under Protective Ventilation.
Acronym: COVAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: P160701; 2016-A01689-42 (Other: IDRCB)
Record Dates: First submitted 2017-09-26; First posted 2017-10-06 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2018-09

CONDITIONS: Acute Respiratory Distress Syndrome; Hypercapnia
Keywords: Extracorporeal CO2 removal (ECCO2-R); ARDS
MeSH Terms: conditions — Respiratory Distress Syndrome; Hypercapnia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Extracorporeal CO2 removal (Other): Extracorporeal CO2 removal (ECCO2-R) (PrismaLung®, Prismaflex ® Baxter)
  Interventions: Device: Extracorporeal CO2 removal (ECCO2-R) (PrismaLung®, Prismaflex ® Baxter)

INTERVENTIONS:
Device: Extracorporeal CO2 removal (ECCO2-R) (PrismaLung®, Prismaflex ® Baxter) — A low-flow CO2 removal device (Prismalung®, Baxter) will be used with a conventional renal replacement therapy (RRT) platform (Prismaflex®, Baxter). In patients already treated with continuous RRT because of renal failure or metabolic acidosis, the HF 1400® (Baxter) set will be used to combine RRT and decarboxylation. Gas flow through the gas exchanger will be set up to 10 L/min, with an oxygen concentration from 0.21 to 1 and a blood flow of 200-400 mL/min. Patients will be ventilated with a target tidal volume of 6 ml/kg (predicted body weight) and a target plateau pressure below 30 cmH2O.

SUMMARY:
Pulmonary vascular dysfunction (DVP) is associated with a pejorative prognosis during ARDS. There is no specific therapeutic intervention to thwart it. Extracorporeal CO2 purification (ECCO2-R) is a technique that has been very rapidly diffused and adopted in intensive care since commercialization of the devices but, the formal clinical evaluation is insufficient. It could significantly improve the prognosis of patients with both DVP and refractory hypercapnia.

DETAILED DESCRIPTION:
This is a prospective, non-comparative, open-label, multicenter regional study, without random drawing or blindfolding.

The primary objective of the study is the correction by ECCO2-R of hypercapnia in patients with DVP in moderate to severe ARDS under protective ventilation.

The primary endpoint is the percentage of patients with hypercapnia correction (defined as a 20% decrease in PaCO2 at H2 of ECCO2-R initiation).

The secondary objectives are:

* Demonstrate that ECCO2-R allows in hypercapnic ARDS and DVP patients to correct hypercapnia with H6 and H24, improve DVP and hemodynamics, reduce alveolar dead space, improvement of respiratory mechanics
* Assess the tolerance of the evaluated technique.

The Secondary endpoints are:

- Relative change of capnia to H6 and H24 in relation to H0; proportion of patients with a decrease of at least 20% of PaCO2 to H6 and H24; changes in echocardiographic indices; hemodynamic parameters; alveolar deadspace and respiratory mechanics to H2, H6 and H24, compared to H0; Complications, Mortality at reanimation discharge (or on D28 if this date occurs before discharge of reanimation).

The intervention is based on the use of ECCO2-R (PrismaLung®, Prismaflex ® Baxter) in eligible patients. ECCO2-R will be initiated as soon as possible after inclusion, for a duration of at least 24 H (possibly prolonged up to 72 H at the decision of reanimator), by jugular or femoral vein-venous.

The size of the catheters, the machine settings, in particular the blood flow and sweep will be standardized according to the state of the art and the recommendations of the manufacturer

The ECO2R venous technique uses devices consisting of a monitor, an exchanger and a pump.

1. The PrismaLung® Kit (Baxter): Single-use EC-marked extracorporeal circuit intended for use for at least 24 hours (maximum 72 hours).

   The PrismaLung® kit is intended for use with the Prismaflex® monitor with software version 8.10 or later and its support in conjunction with Prismaflex® single use treatment sets.
2. The Prismaflex HP-X Set (Baxter): blood line set for extracorporeal blood circulation, EC marked or the HF 1400® set (Baxter) (for extra-corporeal CO2 purification combined with purification).
3. The Prismaflex® monitor (Baxter), EC marked, is used routinely in intensive care (continuous extra-renal purification, therapeutic plasma exchange, haemoperfusion, hemopurification).

So that each center has a dedicated monitor for research, this device will be provided by the Baxter laboratory. The monitor will be equipped with a holder for the Prismalung kit marked CE.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe ARDS according to the Berlin definition;
* Pulmonary vascular dysfunction at echocardiography (pulmonary arterial hypertension, right ventricular dilatation or dyskinesia of the interventricular septum);
* Refractory hypercapnia, defined by a PaCO2 ≥48 mmHg in spite of the reduction of the instrumental dead space and the increase of the respiratory rate.
* Free and informed written consent for persons in a position to consent; consent of the support person/parent/relative in case of incapacity to consent; inclusion in emergency situations (Article L1122-1-2 of the CSP)

Exclusion Criteria:

* Age <18 years;
* Known pregnancy or breastfeeding;
* Contra-indication to curative anticoagulation, thrombocytopenia <50 G / L, heparin-induced thrombocytopenia, known hypersensitivity to heparin or to compounds;
* Femoral or jugular venous access impossible;
* Refractory hypoxemia with indication at ECMO;
* No affiliation to social security or beneficiary

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2018-01-10 (Actual); Primary Completion 2019-02-25 (Actual); Study Completion 2019-03-21 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with corrected hypercapnia | at hour 2 (H2)
  20% decrease in PaCO2 two hours after ECCO2-R initiation

SECONDARY OUTCOMES:
Relative change of capnia at H6 and H24 after ECCO2-R | at hour 6 (H6), at hour 24 (H24)
Proportion of patients with a decrease of at least 20% of PaCO2 to H6 and H24 | H6, H24
Changes in echocardiographic indices | H2, H6, H24
  Changes in echocardiographic indices at H2, H6 and H24
Changes in hemodynamic parameters | H2, H6, H24
  Changes in hemodynamic parameters at H2, H6 and H24
Changes in alveolar deadspace | H2, H6, H24
  Changes in alveolar deadspace at H2, H6 and H24
Changes in respiratory mechanics | H2, H6, H24
  Changes in respiratory mechanics at H2, H6 and H24
Number of complications related to ECCO2-R technique | ICU Discharge or day 28
Percentage of mortality | ICU discharge or day 28

CONTACTS AND LOCATIONS:
Overall Officials: Armand Mekontso Dessap, MD, PhD, Study Chair — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Henri Mondor Hospital, Créteil, France

REFERENCES:
- [Derived] Mekontso Dessap A, Bagate F, Repesse X, Blayau C, Fartoukh M, Canoui-Poitrine F, de Prost N, Vieillard-Baron A. Low-flow ECCO2R conjoined with renal replacement therapy platform to manage pulmonary vascular dysfunction with refractory hypercapnia in ARDS. Heliyon. 2023 Dec 19;10(1):e23878. doi: 10.1016/j.heliyon.2023.e23878. eCollection 2024 Jan 15. PMID 38226285